CLINICAL TRIAL: NCT06602713
Title: Ability of Rotator Cuff Muscle Strength Levels, Assessed by Isokinetic Dynamometry, to Predict Return to Sport After Shoulder Stabilization Surgery by Open Latarjet Procedure
Acronym: ISO-LAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A00418-39
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Latarjet; Shoulder Injuries; Rotator Cuff Injuries
MeSH Terms: conditions — Shoulder Injuries; Rotator Cuff Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: one group of volunteers, one group of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Active Comparator): Questionnaires and exercices
  Interventions: Other: Questionnaires; Other: Exercices
- Patient operated at shoulder by open Latarjet procedure (Experimental): Questionnaires and exercices
  Interventions: Other: Questionnaires; Other: Exercices

INTERVENTIONS:
Other: Questionnaires — Western Ontario Shoulder Instability questionnaire Western Ontario Rotator Cuff questionnaire Shoulder Instability Return to Sport after Injury questionnaire
Other: Exercices — isokinetic evaluation

SUMMARY:
The stabilization surgical treatment by open Latarjet procedure is one of the reference treatments after anterior glenohumeral dislocation in athletes. This surgical technique allows low recurrence rates and high return to sport rates. Indeed, more than 90% of athletes return to sport after this type of surgery, but only 60% are able to resume the same activity as a preinjury level of performance. Therefore, adaptations in the postoperative management of athletes patients seem necessary. Isokinetic dynamometry is considered the gold standard to provide an objective assessment of muscle strength abilities, particularly in the clinical setting. Although rehabilitation exercises are prescribed early after the Latarjet procedure, muscle deconditioning occurs during the postoperative phase, limiting the abilities of the rotator cuff muscles to provide stability to the glenohumeral joint. Therefore, recovery of all components of strength, i.e. maximal strength, power, and strength endurance of the rotator cuff muscles appears crucial for the athletes to return to their sport at the pre-injury level. However, at present, the strength levels to be recovered remain to be defined.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Be aged between 18 and 45
* Occurrence of the injury during the practice of a sporting activity
* Post-traumatic anterior glenohumeral subluxation/dislocation
* Contralateral shoulder with no history of injury
* No other associated shoulder pathology
* Patient scheduled for shoulder stabilizing surgery using an open Latarjet procedure performed by one of the surgeons at the Santy Orthopedic Center (Lyon)
* No contraindication to isokinetic assessment
* Patient having signed informed consent
* Subject affiliated or beneficiary of a social security scheme

Healthy volunteers:

* Be aged between 18 and 45
* Regularly practice a sporting activity
* No contraindication to isokinetic assessment
* Person having signed informed consent
* Subject affiliated or beneficiary of a social security scheme

Exclusion Criteria:

Patient group:

* Contraindication from the sports clinician or surgeon
* Have another pathology in the upper limbs.
* Have constitutional hyperlaxity
* Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Healthy volunteer group (athletes without a history of shoulder pathology):

* Declare a history of pain/injury in the upper limbs in the last 6 months
* Declare a history of orthopedic surgery in the upper limbs
* Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Bilateral glenohumeral rotator muscle strength differences assessed at 4 months postoperatively | 4 months
  Bilateral muscle strength gap at 4 months postoperatively:
  * concentric internal rotators at 60°/s
  * concentric external rotators at 60°/s,
  * eccentric internal rotators at 60°/s,
  * eccentric external rotators at 60°/s,
  * concentric endurance internal rotators at 120°/s,
  * concentric endurance external rotators at 120°/s,
Return to same sport at pre-injury level assessed at 12 months post-operatively | 12 months
  questionnaire to the patient : what sport do you practice, which level?

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France